CLINICAL TRIAL: NCT00463814
Title: A Phase I, Open-Label, Multi-centre Study to Assess the Safety, Tolerability and Pharmacokinetics of a Solid Oral Dosage Formulation (Capsule) of AZD6244 in Patients With Advanced Solid Malignancies
Brief Title: AZD6244 (ARRY-142886) Solid Oral Dosage Formulation in Participants With Advanced Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00005; 2022-500685-10-00 (Registry Identifier: CTIS (EU)); 2006-004497-26 (EudraCT Number)
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Tumor; Cancer
Keywords: Advanced Malignancy; Cancer Eligibility; Malignancy
MeSH Terms: conditions — Neoplasms | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (6):
- Part A: Dose Escalation AZD6244 25 mg (Experimental): Participants will receive a single oral dose of AZD6244 25 mg capsule on Day 1 followed by continuous twice daily (bd) dosing from Day 2 onwards, until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244
- Part A: Dose Escalation AZD6244 50 mg (Experimental): Participants will receive a single oral dose of AZD6244 50 mg capsule on Day 1 followed by continuous dosing from Day 2 onwards, until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244
- Part A: Dose Escalation AZD6244 75 mg (Experimental): Participants will receive a single oral dose of AZD6244 75 mg capsule on Day 1 followed by continuous dosing from Day 2 onwards, until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244
- Part A: Dose Escalation AZD6244 100 mg (Experimental): Participants will receive a single oral dose of AZD6244 100 mg capsule on Day 1 followed by continuous dosing from Day 2 onwards, until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244
- Part B: Relative Bioavailability (Sequence 1) and Safety Assessment Phase (Experimental): Participants in relative bioavailability phase will receive a single oral dose of AZD6244 100 mg free-base suspension (mix and drink) on Day 1. Following a washout period of 7 days, participants will receive a single oral dose of AZD6244 75 mg capsule on Day 8 (Sequence 1). In the safety assessment phase, participants who will participate in the relative bioavailability phase will receive oral AZD6244 75 mg capsule bd dosing from Day 9 onwards until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244
- Part B: Relative Bioavailability (Sequence 2) and Safety Assessment Phase (Experimental): Participants in relative bioavailability phase will receive a single oral dose of AZD6244 75 mg capsule on Day 1. Following a washout period of 7 days, participants will receive a single oral dose of AZD6244 100 mg free-base suspension (mix and drink) on Day 8 (Sequence 2). In the safety assessment phase, participants who will participate in the relative bioavailability phase will receive oral AZD6244 75 mg capsule bd dosing from Day 9 onwards until disease progression or another protocol-defined discontinuation criterion will be met, whichever will occur first.
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — Participants will receive single oral dose of AZD6244 as described in arm description.
  Other Names: ARRY-142886

SUMMARY:
The primary purpose of the study is to assess the safety, tolerability and pharmacokinetics of a capsule of AZD6244 in participants with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* cancer which is refractory to standard therapies
* World Health Organization (WHO) performance status 0 to 2
* evidence of post-menopausal status or negative pregnancy test

Exclusion Criteria:

* Radiotherapy/chemotherapy within 21 days prior to entry
* brain metastases/spinal cord compression unless stable off steroids/anticonvulsants
* evidence of severe/uncontrolled systemic disease
* participated in an investigational drug study within 30 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-03-08 (Actual); Primary Completion 2008-06-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) in Part A and Part B | Day 1 through 11.8 months (maximum observed duration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Part A and Part B | Day 1 through 11.8 months (maximum observed duration)
  Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of hematology, clinical chemistry, and urinalysis.
Number of Participants With Abnormal Vital Signs Reported as TEAEs in Part A and Part B | Day 1 through 11.8 months (maximum observed duration)
  Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (blood pressure, oxygen saturation, weight, and pulse rate).
Number of Participants With Abnormal Echocardiogram (ECHO) Parameters Reported as TEAEs in Part A and Part B | Day 1 through 11.8 months (maximum observed duration)
  Number of participants with abnormal ECHO parameters reported as TEAEs are reported.
Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs in Part A and Part B | Day 1 through 11.8 months (maximum observed duration)
  Number of participants with abnormal ECG parameters reported as TEAEs are reported.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Cmax of AZD6244 in Part A is reported.
Cmax of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Cmax of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC of AZD6244 in Part A is reported.
Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post Dose (AUC[0-12]) of AZD6244 (Part A) | Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The AUC(0-12) of AZD6244 in Part A is reported.
AUC of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Post Dose (AUC[0-24]) of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC(0-24) of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Time to Reach Maximum Plasma Concentration (Tmax) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Tmax of AZD6244 in Part A is reported.
Tmax of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Tmax of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Half-life (t1/2) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The t1/2 of AZD6244 in Part A is reported.
t1/2 of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The t1/2 of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Total Apparent Drug Clearance (CL/F) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The CL/F of AZD6244 in Part A is reported.
CL/F of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The CL/F of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Volume of Distribution at Steady State (Vss/F) of AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Vss/F of AZD6244 in Part A is reported.
Vss/F of AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Vss/F of AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Cmax of N-desmethyl AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Cmax of N-desmethyl AZD6244 in Part A is reported.
Cmax of N-desmethyl AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Cmax of N-desmethyl AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
AUC of N-desmethyl AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC of N-desmethyl AZD6244 in Part A is reported.
AUC(0-12) of N-desmethyl AZD6244 (Part A) | Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The AUC(0-12) of N-desmethyl AZD6244 in Part A is reported.
AUC of N-desmethyl AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC of N-desmethyl AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
AUC(0-24) of N-desmethyl AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC(0-24) of N-desmethyl AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Tmax of N-desmethyl AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Tmax of N-desmethyl AZD6244 in Part A is reported.
Tmax of N-desmethyl AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Tmax of N-desmethyl AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
t1/2 of N-desmethyl AZD6244 (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The t1/2 of N-desmethyl AZD6244 in Part A is reported.
t1/2 of N-desmethyl AZD6244 (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The t1/2 of N-desmethyl AZD6244 in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Cmax of AZD6244 Amide (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Cmax of AZD6244 amide in Part A is reported.
Cmax of AZD6244 Amide (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Cmax of AZD6244 amide in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
AUC(0-12) of AZD6244 Amide (Part A) | Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The AUC(0-12) of AZD6244 amide in Part A is reported.
Area Under the Plasma Concentration-time Curve From Time Zero to 4 Hours Post Dose (AUC[0-4]) of AZD6244 Amide (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC(0-4) of AZD6244 amide in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
AUC(0-24) of AZD6244 Amide (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The AUC(0-24) of AZD6244 amide in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Tmax of AZD6244 Amide (Part A) | Day 1: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose; Day 8: Pre-dose (within 10 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, and 12 hours post-dose
  The Tmax of AZD6244 amide in Part A is reported.
Tmax of AZD6244 Amide (Part B Single Dose) | Days 1 and 8: Pre-dose (within 30 minutes of dosing); 5, 15, and 30 minutes, 1, 1.5, 2, 4, 8, 12, and 24 hours post-dose
  The Tmax of AZD6244 amide in Part B is reported. Day 1 and Day 8 in Part B are the first days of two periods in crossover bioavailability assessment of two AZD6244 formulations: capsule versus the free-base suspension.
Cmax of AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Cmax of AZD6244 in Part B is reported.
Tmax of AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Tmax of AZD6244 in Part B is reported.
AUC(0-4) of AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-4) of AZD6244 in Part B is reported.
Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC[0-t]) of AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-t) of AZD6244 in Part B is reported.
Cmax of N-desmethyl AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Cmax of N-desmethyl AZD6244 in Part B is reported.
Tmax of N-desmethyl AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Tmax of N-desmethyl AZD6244 in Part B is reported.
AUC(0-4) of N-desmethyl AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-4) of N-desmethyl AZD6244 in Part B is reported.
AUC(0-t) of N-desmethyl AZD6244 (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-t) of N-desmethyl AZD6244 in Part B is reported.
Cmax of AZD6244 Amide (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Cmax of AZD6244 amide in Part B is reported.
Tmax of AZD6244 Amide (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The Tmax of AZD6244 amide in Part B is reported.
AUC(0-4) of AZD6244 Amide (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-4) of AZD6244 amide in Part B is reported.
AUC(0-t) of AZD6244 Amide (Part B Multiple Doses) | Days 15 and 22: Pre-dose (within 10 minutes of dosing); 1, 2, and 4 hours post-dose
  The AUC(0-t) of AZD6244 amide in Part B is reported.
Percentage Inhibition of Extracellular Signal-regulated Kinase (ERK) Phosphorylation | 1, 4, 8, and 24 hours post-dose on Day 1 (Part A and Part B) and Day 8 (Part B)
  Percentage inhibition of ERK phosphorylation is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (4):
- Research Site, Aurora, Colorado, United States
- Netherlands (2):
  - Research Site, Nijmegen
  - Research Site, Utrecht
- Research Site, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Boers-Sonderen MJ, Desar IM, Blokx W, Timmer-Bonte JN, van Herpen CM. A prolonged complete response in a patient with BRAF-mutated melanoma stage IV treated with the MEK1/2 inhibitor selumetinib (AZD6244). Anticancer Drugs. 2012 Aug;23(7):761-4. doi: 10.1097/CAD.0b013e328350737d. PMID 22293660
- See also: CSR_redacted_2023 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1532C00005&attachmentIdentifier=719057c6-d08a-4048-8598-9a0028c402fb&fileName=D1532C00005__CSRStudy_Synopsis_Redacted.pdf&versionIdentifier=